CLINICAL TRIAL: NCT03410004
Title: Study of Chidamide as a Single-agent Treatment for Patients With Relapse or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) and Follicular Lymphoma (FL)
Brief Title: Chidamide for Patients With Relapse or Refractory Diffuse Large B-Cell Lymphoma and Follicular Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, vice president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-B07
Record Dates: First submitted 2018-01-12; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Experimental
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Drug: Chidamide 30mg orally BIW. Treatment cycles are repeated every 4 weeks.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide 30mg orally BIW. Treatment cycles are repeated every 4 weeks.
  Other Names: Chidamide single agnet

SUMMARY:
Study of Chidamide as a single-agent treatment for patients with relapse or refractory Diffuse Large B-Cell Lymphoma (DLBCL) and Follicular Lymphoma (FL)

DETAILED DESCRIPTION:
Chidamide，a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. The aim of this study was to observe the efficacy and safety of Chidamide as a single-agent treatment in patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) and Follicular Lymphoma (FL). Moreover, the aim was to study the correlation of clinical efficacy to mutation of certain genes as well.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as Diffuse Large B-Cell Lymphoma (DLBCL) and Follicular Lymphoma (FL) according to "2016 WHO classification of tumors of haematopoietic and lymphoid tissues";
2. Patients must have received systemic treatment (including chemotherapy or Hematopoietic stem cell transplantation), but did not achieve remission or had relapse after remission;
3. At least one measurable lesion;
4. Age 18-75 years, male or female;
5. ECOG performance status 0-1;
6. Without bone marrow involvement. Blood routine test: absolute neutrophil count ≥1.5 × 109/L, platelet ≥80 × 109/L, Hb ≥ 90g/L;.
7. Life expectancy no less than 3 months;
8. Not received chemotherapy, targeted medicine or stem cell transplantation 3 weeks before enrollment;
9. Patients have signed the Informed Consent Form.

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures.
2. QTc elongation with clinical significance ( male˃ 450ms, female˃ 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment;
3. pericardial effusion ≥10mm sum of echo-free spaces by echocardiography;
4. Patients have undergone organ transplantation;
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment.
6. Patients with active hemorrhage.
7. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction.
8. Patients with active infection, or with continuous fever within 14 days prior to enrollment.
9. Had major organ surgery within 6 weeks prior to enrollment.
10. Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum).
11. Patients with mental disorders or those do not have the ability to consent.
12. Patients with drug abuse, long term alcoholism that may impact the results of the trial.
13. Patients who have central nervous system involvements;
14. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-25 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | up to 2 years
  the total proportion of patients with complete response（CR or CRu）and partial response（PR）

SECONDARY OUTCOMES:
Disease Control Rate （DCR） | up to 2 years
  the total proportion of patients with complete response（CR or CRu）, partial response（PR）and Stable Disease（SD）
progression-free survival（PFS） | 2 years
  Time from treatment until disease progression or death
overall survival（OS） | 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Dr., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No